CLINICAL TRIAL: NCT00940199
Title: Prospective Randomized Trial of Standard Versus pH-adjusted Radiocolloid for Patients Undergoing Sentinel Lymph Node Mapping and Biopsy for Breast Cancer PASSION - P Trial: Ph Adjusted Sulfur-Colloid, Sentinel Initiative ON Pain Trial
Brief Title: PASSION - P Trial: Ph Adjusted Sulfur-Colloid, Sentinel Initiative ON Pain Trial
Acronym: PassionP
Status: Completed | Type: Observational
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: COL Alexander Stojadinovic, Walter Reed Army Medical Center
Other Study IDs: WU#06-20027; WU#06-20027
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer, sentinel lymph node mapping, biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Standard of Care: I:Application of L-M-X topical anesthetic cream 4% to the breast within one hour of sub-areaolar injection of 4 ml 99mTc-sulfur colloid (1 mCi in normal saline)
- 1 mCi in sodium bicarbonate: II. Sub-areolar injection of 4 ml pH-adjusted 99mTc-sulfur colloid (1 mCi in sodium bicarbonate)
- 1 mCi in 1% Lidocaine: III. Sub-areolar injection of 4 ml pH-adjusted 99mTc-sulfur colloid (1 mCi in 1% Lidocaine)
- 1 mCi in sodium bicarbonate + 1% Lidocaine: IV. Sub-areolar injection of 4 ml pH-adjusted 99mTc-sulfur colloid (1 mCi in sodium bicarbonate + 1% Lidocaine)

SUMMARY:
Patients with breast cancer scheduled to undergo sentinel lymph node mapping and biopsy will be randomly assigned to one of four treatment groups:

I: (Standard of Care at WRAMC): Application of L-M-X topical anesthetic cream 4% to the breast within one hour of sub-areaolar injection of 4 ml 99mTc-sulfur colloid (1 mCi in normal saline)

II. Sub-areolar injection of 4 ml pH-adjusted 99mTc-sulfur colloid (1 mCi in sodium bicarbonate)

III. Sub-areolar injection of 4 ml pH-adjusted 99mTc-sulfur colloid (1 mCi in 1% Lidocaine)

IV. Sub-areolar injection of 4 ml pH-adjusted 99mTc-sulfur colloid (1 mCi in sodium bicarbonate + 1% Lidocaine)

The primary study outcome is pain, which will be evaluated for each study group before, and after radiocolloid injection utilizing a standardized 10-point Likert scale, the Wong-Baker FACES Pain Rating Scale, and the McGill Pain Questionnaire. Physician appraisal of patient pain (Wong-Baker FACES Pain Rating Scale) will be estimated during the radiocolloid injection and compared with that of the patient.

DETAILED DESCRIPTION:
Null hypothesis: There is no difference in overall pain intensity between standard and pH adjusted radiocolloid for patients undergoing sentinel lymph node mapping and biopsy for breast cancer.

Objectives and scientific aims:

To compare the intensity of pain (Wong-Baker FACES Pain Rating Scale + McGill Pain Questionnaire) associated with WRAMC's current standard and pH-adjusted radiocolloid for patients undergoing sentinel lymph node mapping and biopsy for breast cancer.

To assess objectively physician appraisal of patient pain during the radiocolloid injection and compare physician interpreted pain score with patient reported pain score.

Define the success rate of intra-operative SLN identification for each study group.

ELIGIBILITY:
Inclusion criteria:

1. Female military healthcare beneficiaries should be over 18 years of age and capable of providing informed consent indicating awareness of the investigational nature of this trial, in keeping with institutional policy.
2. Written informed consent must be obtained from each patient prior to entering the study.
3. Female military healthcare beneficiaries with early breast cancer scheduled to undergo sentinel lymph node mapping and biopsy at WRAMC

Exclusion criteria:

1. Female military healthcare beneficiaries with chronic pain syndrome (e.g. fibromyalgia) undergoing active narcotic-based treatment.
2. Female military healthcare beneficiaries participating in other clinical trials the requirements of which may preclude complete involvement in this study.
3. Female military healthcare beneficiaries with significant allergy to local anesthetics.
4. Female military healthcare beneficiaries presenting with large (>4cm), clinically node positive, painful, locally advanced breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of female military health care beneficiaries over the age of 18 years presenting with the diagnosis of breast cancer who meet inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To compare the intensity of pain (Wong-Baker FACES Pain Rating Scale + McGill Pain Questionnaire) associated with WRAMC's current standard and pH-adjusted radiocolloid for patients undergoing sentinel lymph node mapping and biopsy for breast cancer. | June 2009

SECONDARY OUTCOMES:
To assess objectively physician appraisal of patient pain during the radiocolloid injection and compare physician interpreted pain score with patient reported pain score | June 2009

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stojadinovic, M.D., Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Stojadinovic A, Peoples GE, Jurgens JS, Howard RS, Schuyler B, Kwon KH, Henry LR, Shriver CD, Buckenmaier CC. Standard versus pH-adjusted and lidocaine supplemented radiocolloid for patients undergoing sentinel-lymph-node mapping and biopsy for early breast cancer (PASSION-P trial): a double-blind, randomised controlled trial. Lancet Oncol. 2009 Sep;10(9):849-54. doi: 10.1016/S1470-2045(09)70194-9. Epub 2009 Aug 5. PMID 19664956